CLINICAL TRIAL: NCT03966547
Title: Changes in Cerebral Blood Flow (CBF) in Prone and Sitting Position Before and After GSP-block and Before and After Epidural Blood-patch: A Substudy of NCT03652714
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Main study concluded before enrollment
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Responsible Party: Principal Investigator, Mads Seit Jespersen, Medical Doctor, Primary Investigator, University Hospital Bispebjerg and Frederiksberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: GSPB-2018-SUB
Record Dates: First submitted 2019-05-14; First posted 2019-05-29 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Postdural Puncture Headache; Sphenopalatine Ganglion Block
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Local anesthetic (Experimental)
  Interventions: Procedure: Ganglion sphenopalatine block with local anesthetic administered on study GSPB-2018
- Isotonic NaCl (Placebo Comparator)
  Interventions: Procedure: Ganglion sphenopalatine block with placebo administered on study GSPB-2018

INTERVENTIONS:
Procedure: Ganglion sphenopalatine block with local anesthetic administered on study GSPB-2018 — Block performed with bilaterally inserted q-tips with 1:1 mixture of lidocaine 40mg/ml and ropivacaine 5mg/mL as per GSPB-2018.
  Arms: Local anesthetic
Procedure: Ganglion sphenopalatine block with placebo administered on study GSPB-2018 — Block performed with bilaterally inserted q-tips with isotone NaCl as per GSPB-2018.
  Arms: Isotonic NaCl

SUMMARY:
The purpose of this optional sub-study to GSPB-2018 (NCT03652714) is to evaluate the changes in cerebral blood flow (CBF) under different conditions to understand if postdural puncture headache is caused by changes in the cerebral blood flow and if treatment normalises that change.

ELIGIBILITY:
Study Population:

Subjects who have consented to participate in GSPB-2018 will be approached for participation in this sub-study. Subjects who have consented to participate in GSPB-2018 are not required to participate in this sub-study.

Inclusion Criteria:

* Age > 18 years
* Patients with postdural puncture headache defined as moderate to severe postural headache (VAS >= 30mm) after lumbar puncture or accidental dural puncture during epidural insertion with an onset within 3 days following the puncture.
* Lack of headache remission within 1 day after dural puncture and after treatment with fluids, caffeine and paracetamol
* Patients who have given their written informed consent for participation in the study and substudy after fully understanding the protocol content and limitations.

Exclusion Criteria:

* Patients who cannot cooperate to the study
* Patients who does not understand or speak Danish
* Allergy to the drugs used in the study
* Has taken opioids within 12 hours prior to intervention
* No possible transcranial window on transcranial doppler. If not possible to find a useable window to get measurement the patient will be excluded and replaced with another patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change in Cerebral Blood Flow velcity (CBF) in supine versus upright position compared to effect of treatment. | <1h before and 1 hour after each intervention
  Change in mean, minimum and maximum Cerebral Blood Flow velcity in cm/sec (CBF) in supine versus upright position compared to effect of treatment.
Comparison of paint rating (0-100 on a visual analogue scale, VAS) and Cerebral Blood Flow velocity (CBF) before and after each intervention. | <1h before and 1 hour after each intervention
  Pain intensity measured with a pain rating (0-100mm on a visual analogue scale, VAS) in supine position and as worst experienced pain after the patient has been upright for 30 seconds or the worst experienced pain while attempting to stand if the rating has to be interrupted.
  Cerebral Blood Flow velocity (CBF) measured as mean blood flow in cm/sec.

SECONDARY OUTCOMES:
Change in Cerebral Blood Flow velocity (CBF) in supine position before and after interventions. | <1h before and 1 hour after each intervention
  Changes in mean, minimum and maximum Cerebral Blood Flow velocity in cm/sec (CBF) before and after treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Bispebjerg and Frederiksberg Hospital, University of Copenhagen, Copenhagen
  - Rigshospitalet, University of Copenhagen, Copenhagen